**Title:** High-intensity Inspiratory Muscle Training as a Pre-cardiac Rehabilitation in Heart

Disease

NCT Number: NCT06127147

**Date:** 12/12/2023

## **Statistical Analysis Plan**

Statistical analyses will be performed using SPSS version 21.0 (IBM, Armonk, NY). The Shapiro–Wilk test will be used to evaluate normality of the data distribution for each variable. The continuous variables will be reported as mean 6 SD, and the categorical variables will be presented in absolute frequencies and percentages. Nominal data will be compared using a Chi-square test. For comparison between the baseline and postintervention, the paired-samples t test or Mann–Whitney U test will be applied based on normality distribution. Change from the baseline values will also be calculated as the mean difference for each measure. Treatment effect and between-group comparisons will be evaluated based on mean differences using analysis of variance. Effect sizes will be provided as eta square, which are interpreted as small effect (0.01), medium effect (0.06), and large effect (0.14). The alpha value will be set at alpha = 0.05 for all outcomes.